CLINICAL TRIAL: NCT02779491
Title: Evaluation of a 5-a-day Fruit and Vegetable Mobile Phone Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REC10186
Record Dates: First submitted 2016-04-13; First posted 2016-05-20 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Nutritional Status; Nutrition Assessment
Keywords: fruit and vegetables; food intake; knowledge

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intervention for two weeks (Experimental): Receipt of the mobile phone application for two weeks
  Interventions: Behavioral: 5-a-day fruit and vegetable mobile phone application
- Control for two weeks (No Intervention): Usual habitual activity - no receipt of mobile phone application for two weeks
- Intervention for four weeks (Experimental): Receipt of the mobile phone application for four weeks
  Interventions: Behavioral: 5-a-day fruit and vegetable mobile phone application
- Control for four weeks (No Intervention): Usual habitual activity - no receipt of mobile phone application for two weeks

INTERVENTIONS:
Behavioral: 5-a-day fruit and vegetable mobile phone application — 5-a-day fruit and vegetable mobile phone application
  Arms: Intervention for four weeks; Intervention for two weeks

SUMMARY:
This is a randomized controlled trial to assess the impact of a novel fruit and vegetable mobile phone application on fruit and vegetable intakes, knowledge and attitudes.

DETAILED DESCRIPTION:
The 5-a-day fruit and vegetable (FV) message from the WHO recommends consumption of five 80g portions of different FV per day for health reasons. Recent research suggests that the details of the message are poorly understood by the population as a whole, by low consumers of FV and by those in demographic groups of traditional low FV consumption, and that this poor knowledge impacts on implementation of the message to result in low FV intakes. To aid implementation of the recommendations, investigators have developed a 5-a-day FV mobile phone application (app) prototype. The basic prototype app will provide information on the 5-a-day message, allow users to input consumption, and provides consumers with accurate knowledge of their adherence to the recommendations. This study will investigate the use and impact of the prototype app on FV intakes over a two or four week period. For significant impacts on health, sustained user engagement and use will be required. Up to 100 participants will be randomised to either receive or not receive the app, and will be asked to use the app for the following two or four weeks. FV intake will be assessed at baseline, 2 weeks, 4 weeks. Measures of app use will also be taken at these time points. Measures of FV knowledge will also be measured at these time points. Measures of FV attitudes were initially planned but not undertaken to reduce demand characteristics for participants. The investigators anticipate that changes in intakes will be mediated by changes in knowledge and attitudes.

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent
* speaks English, owns an android mobile telephone
* able and willing to use phone and complete all measures

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-30 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
Data will be available from the PI on request
Time Frame: Following publication of findings in a peer-reviewed journal article.
Access Criteria: Reasonable request of the PI.

REFERENCES:
- [Derived] Appleton KM, Passmore D, Burn I, Pidgeon H, Nation P, Boobyer C, Jiang N. An Interactive Mobile Phone App (SMART 5-A-DAY) for Increasing Knowledge of and Adherence to Fruit and Vegetable Recommendations: Development and Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Nov 20;7(11):e14380. doi: 10.2196/14380. PMID 31746766

RESULTS

PARTICIPANT FLOW:
Groups:
- Control for Four Weeks: Usual habitual activity - no receipt of mobile phone application for four weeks
Period: Overall Study
Arm/Group | Intervention for Two Weeks | Control for Two Weeks | Intervention for Four Weeks | Control for Four Weeks
Started | 32 | 27 | 18 | 17
Completed | 32 | 26 | 17 | 15
Not Completed | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention for Two Weeks | Control for Two Weeks | Intervention for Four Weeks | Control for Four Weeks | Total
Number analyzed (Participants) | 32 | 27 | 18 | 17 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.3 (7.7) | 21.4 (5.3) | 25.9 (7.9) | 25.9 (7.9) | 23.4 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 12 | 12 | 63
  Male | 10 | 10 | 6 | 5 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 32 | 27 | 18 | 17 | 94
FV intake [Mean (Standard Deviation); unit: FV portions per day] | 3.9 (1.5) | 3.7 (2.3) | 4.4 (1.2) | 3.7 (1.3) | 3.9 (1.9)
FV knowledge [Mean (Standard Deviation); unit: Scores on a scale] — FV knowledge will be assessed by the FV knowledge questionnaire published in Appleton et al. J Hum Nutr Diet, 2018;31:121-130. The questionnaire assesses four aspects of FV knowledge in relation to the UK 5-a-day recommendations. Scores are provided for the subscale for portion sizes, where positive scores are given for correct responses, and negative scores for incorrect responses. Min. max scores are -27, 27. Higher scores show greater knowledge.
  Scores on a scale | -5.5 (6.5) | -7.6 (6.3) | -8.2 (5.1) | -8.1 (4.8) | -7.1 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Fruit and Vegetable Intakes (Self-report, Questionnaire Assessment)
Description: Self-report, questionnaire assessment
Time Frame: Intervention end
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: FV portions per day
Arm/Group | Intervention for Two Weeks | Control for Two Weeks | Intervention for Four Weeks | Control for Four Weeks
Number analyzed (Participants) | 32 | 27 | 18 | 17
FV portions per day | 3.8 (1.7) | 2.6 (2.0) | 5.2 (1.6) | 4.0 (1.8)

2. Secondary Outcome: Fruit and Vegetable Knowledge (Questionnaire Assessment)
Description: FV knowledge will be assessed by the FV knowledge questionnaire published in Appleton et al. J Hum Nutr Diet, 2018;31:121-130. The questionnaire assessed four aspects of FV knowledge in relation to the UK 5-a-day recommendations. The portion sizes subscale is provided, where positive scores are given for correct responses, and negative scores for incorrect responses. Min. max scores are -27, 27. Higher scores show greater knowledge.
Time Frame: Intervention end
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention for Two Weeks | Control for Two Weeks | Intervention for Four Weeks | Control for Four Weeks
Number analyzed (Participants) | 32 | 27 | 18 | 17
scores on a scale | -2.5 (7.7) | -5.5 (8.7) | -7.7 (9.5) | -5.3 (8.1)

3. Secondary Outcome: App Usage
Description: Number of days on which users interacted with the app.
Time Frame: Intervention end
Population: Control participants did not receive the app, so no app data is available
Measure: Mean (Standard Deviation); unit: days used
Arm/Group | Intervention for Two Weeks | Control for Two Weeks | Intervention for Four Weeks | Control for Four Weeks
Number analyzed (Participants) | 32 | 0 | 18 | 0
days used | 11.4 (7.2) |  | 13.7 (9.2) |

ADVERSE EVENTS:
Time Frame: Study duration - 2 or 4 weeks, as defined at study entry.
Description: Questions from researcher
Arm/Group | Intervention for Two Weeks | Control for Two Weeks | Intervention for Four Weeks | Control for Four Weeks
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/27 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/27 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/32 | 0/27 | 0/18 | 0/17

LIMITATIONS AND CAVEATS:
Assessment of FV attitudes was originally planned but were not measured in the actual study to reduce demand characteristics for participants considering the large number of existing measures related to FV. No data on FV attitudes were collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT02779491/Prot_SAP_000.pdf